CLINICAL TRIAL: NCT06833931
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study of PGN-EDO51 With a Long-Term Extension in Participants With Duchenne Muscular Dystrophy Amenable to Exon 51-Skipping Treatment (CONNECT2-EDO51)
Brief Title: A Study of PGN-EDO51 or Placebo in People With Duchenne Muscular Dystrophy Amenable to Exon 51-Skipping Treatment
Acronym: CONNECT2-EDO51
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Global PGN-EDO51 development voluntarily discontinued by Sponsor
Sponsor: PepGen Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PGN-EDO51-103; U1111-1303-9370 (Other: WHO); 2023-508383-29-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: Enhanced Delivery Oligonucleotide; Peptide-conjugated phosphorodiamidate; Morpholino oligomer; Oligonucleotide; Exon 51; Next-generation oligonucleotide; Cell-penetrating peptide; Muscular Dystrophies; Neuromuscular Disease; Dystrophin production; Splice correcting oligonucleotide; Endosomal Escape; Delivery to the cell nucleus; Antisense oligonucleotide; phosphorodiamidate morpholino oligomer (PPMO)
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies; Neuromuscular Diseases | interventions — Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PGN-EDO51 at Dose Level 1 or Placebo every 4 weeks (Experimental)
  Interventions: Drug: IV infusion; Other: Placebo
- PGN-EDO51 at Dose Level 2 or Placebo every 4 weeks (Experimental)
  Interventions: Drug: IV infusion; Other: Placebo

INTERVENTIONS:
Drug: IV infusion — IV infusion
Other: Placebo — IV infusion

SUMMARY:
The study consists of 3 periods: A Screening Period (up to 45 days), a double-blind, placebo-controlled Multiple Ascending Dose (MAD) Period (28 weeks), and a Long-Term Extension (LTE) Period (108 weeks).

The primary purpose of the MAD period is to evaluate the safety and tolerability and levels of dystrophin after multiple ascending intravenous (IV) doses of PGN-EDO51 administered to participants with Duchenne muscular dystrophy (DMD). During the MAD period, participants will be randomized to either receive PGN-EDO51 or placebo in a 3:1 fashion, meaning that participants have a 75% chance of receiving PGN-EDO51 and a 25% chance of receiving placebo during this period. The primary purpose of the open-label LTE period is to evaluate the long-term safety and tolerability of PGN-EDO51 in participants who have completed the MAD period. All participants who roll-over into the LTE will receive PGN-EDO51 (no placebo in the LTE).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of DMD with a genetic alteration that can be treated by skipping exon 51
* Body weight at least 25kg (55lbs)
* Performance of Upper Limb (PUL) 2.0 entry score of at least 4

Exclusion Criteria:

* Known history or presence of any clinically significant conditions that may interfere with study safety assessments
* Treatment with any gene replacement therapy for the treatment of DMD at any time
* Current or recent systemic infection within 2 weeks prior to Screening or infection requiring IV antibiotics within 4 weeks prior to Screening
* Recent surgery requiring anesthesia within 3 months prior to Screening or expected surgery requiring general anesthesia during the study

Ages: 6 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events (safety and tolerability of PGN-EDO51 during the MAD period) | Signing of informed consent to Week 28
Dystrophin levels (MAD period) | Baseline to Week 28
Adverse events and serious adverse events (safety and tolerability of PGN-EDO51 during the LTE period) | Signing of informed consent to Week 108

SECONDARY OUTCOMES:
Plasma pharmacokinetic (PK) parameters (MAD period) | Baseline to Week 28
  Maximum observed plasma concentration of PGN-EDO51
Plasma pharmacokinetic (PK) parameters (MAD period) | Baseline to Week 28
  Time to maximum observed plasma concentration of PGN-EDO51
Plasma pharmacokinetic (PK) parameters (MAD period) | Baseline to Week 28
  Apparent terminal half-life of PGN-EDO51
Plasma pharmacokinetic (PK) parameters (MAD period) | Baseline to Week 28
  Area under the curve for concentration time of PGN-EDO51
Skeletal muscle concentration of PGN-EDO51 (MAD period) | Baseline to Week 28
  Change from baseline in skeletal muscle concentration of PGN-EDO51 after multiple doses
Plasma pharmacokinetic (PK) parameters (LTE period) | Baseline to Week 104
  PK sampling for PGN-EDO51 and PGN-PMO51 plasma levels